CLINICAL TRIAL: NCT03802877
Title: ACTIVating and Engaging PAtients Through Clinical Interaction Redesign and Electronically- Integrated Novel Technologies Gestational Diabetes
Brief Title: Active Patient GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Principal Investigator, Kaberi Dasgupta, MD, MSc, FRCP (C), Associate Professor of Medicine, McGill University; Physician Scientist and Director, Centre for Outcomes Research and Evaluation (CORE), Research Institute of the McGill University Health Centre (RI-MUHC), McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: GRT 2017-16
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes
Keywords: gestational weight gain; large for gestational age status; step counts; physical activity; health coaching; ePlatform; pedometer
MeSH Terms: conditions — Diabetes, Gestational; Gestational Weight Gain; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a feasibility (pilot) interventional study with a factorial design
Masking Description: This is a behavioural intervention study. The participant, care provider, and investigator cannot be masked. Outcomes being assessed are objective (weight, steps, etc.) or are participant perspectives that preclude masking. Allocation is concealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Resource bank (Active Comparator): The web-based resource bank includes information and perspectives about GDM, nutrition, and physical activity. The information is presented through video capsules, on-line text, printable pdfs, and podcasts. It is presented by health care professionals and patients.
  Interventions: Behavioral: Resource bank
- Resource bank and ePlatform (Experimental): In addition to resource bank access, participants will receive a digital scale, physical activity monitor (pedometer), and ePlatform log-in information. They will track daily weights and step counts. They will receive prompts to access educational and motivational tools based on the data that they enter and whether or not they enter data. The investigators will use the ePlatform developed by StepsCount, a Canadian pedometer company with a well-developed ePlatform for pedometer data upload, tracking, and automated messaging. The company is permitting us further customization for study purposes. Data will be uploaded onto a secure cloud-based platform controlled by the pedometer and digital scale companies.
  Interventions: Behavioral: Resource bank; Behavioral: ePlatform
- Resource bank and health coach (Experimental): In addition to resource bank access, the coach will contact the participant weekly (telephone, text, email) to discuss progress and challenges in terms of achieving physical activity goals, rate of GWG, and maintaining health eating patterns, as well as any concerns.Participants not randomized to a coaching strategy will be advised to consult with their treating healthcare team directly if they develop symptoms of concern.
  The coach will encourage participants to track their weight gain and physical activity (e.g., walks, classes, activity lists, etc.) and to share this information. However, they will not have access to the study ePlatform and will not be provided with pedometers or digital scales.
  Interventions: Behavioral: Resource bank; Behavioral: Health coach
- Resource bank with ePlatform and coach (Experimental): Participants will have resource bank access as well as ePlatform and coaching interventions.The health coach will have access to the data on the ePlatform. They will receive telephone calls from the research assistant/health coach if they are off target despite the platform tools and support. They will be encouraged to consult the resource bank and will brainstorm with the health coach to decide how to achieve their GWG and step count targets.
  Interventions: Behavioral: Resource bank; Behavioral: ePlatform; Behavioral: Health coach

INTERVENTIONS:
Behavioral: Resource bank — See intervention arm descriptions
Behavioral: ePlatform — See intervention arm descriptions
  Arms: Resource bank and ePlatform; Resource bank with ePlatform and coach
Behavioral: Health coach — See intervention arm descriptions
  Arms: Resource bank and health coach; Resource bank with ePlatform and coach

SUMMARY:
Among women with GDM, the investigators will determine if a strategy of (1) a website-based information and motivational resource bank; (2) biosensor/ePlatform-based physical activity and GWG tracking; and/or (3) a health coach will lead to more favourably outcomes; namely, GWG closer to target, higher physical activity levels, better glycemic and blood pressure control, and lower incidence of LGA in offspring.

The current project is designed to assess feasibility and usability to inform the development of a large randomized controlled trial. The investigators will monitor the implementation process and examine patient-oriented outcomes, including perceptions of utility, challenges, and burden. These will be assessed through telephone-based in-depth interview.

Methodology / Study design This is a feasibility randomized controlled trial with a factorial design. The investigators will recruit women with a diagnosis of GDM between 20 and less than 32 weeks' pregnancy. All will receive access to a website resource bank with tips and resources to optimize physical activity and dietary intake a quality during pregnancy. In addition, they will be randomized to one of the four following groups: (1) No additional intervention; (2) ePlatform-based automated support combined with pedometer-based physical activity monitoring and digital scale-based weight monitoring; (3) weekly telephone calls with a health coach to discuss physical activity, eating, gestational weight gain; (4) combination of ePlatform and telephone calls from a health coach.

The investigators will evaluate recruitment rates, drop-out rates, women's perceptions of the strengths and limitations of the strategy, and ease and feasibility of outcome assessment. Assessments will be through in-clinic assessments, on-line questionnaires, clinic-based measures, mailed-in pedometers, and telephone-based interviews. Assessments will be at study entry and two to three weeks before the expected date of delivery or date of scheduled C-section. There will be a telephone-based interview at 12 weeks postpartum.

DETAILED DESCRIPTION:
Our overarching aim is to determine, among women with gestational diabetes (GDM), if a strategy of (1) a website-based information and motivational resource bank; (2) biosensor/ePlatform-based physical activity and gestational weight gain (GWG) tracking; and/or (3) a health coach will lead to more favourable outcomes; namely, GWG closer to target, higher physical activity levels, better glycemic and blood pressure control, and lower incidence of large for gestational age (LGA) in offspring.

The current project is designed to assess feasibility and usability to inform the development of a large randomized controlled trial. The specific aims of this feasibility study are:

1. To determine the proportion of candidates with GDM who accept to participate in the study at each site (recruitment rates); a minimum overall average recruitment rate of 25/month would favour proceeding to a larger trial.
2. To evaluate participant use (log ins) and perceived utility (interviews) of the website resource that the investigators are developing; a minimum average of 5 log-ins overall would favour proceeding to a larger trial
3. To determine use (number of planned weekly conversations completed) and perceived utility (interviews) of the health coaching intervention; a minimum completion of 50% of the planned weekly conversations would favour retaining this treatment arm in a larger trial
4. To determine use (data upload of step counts and weight data onto ePlatform) and perceived utility (interviews) of the ePlatform intervention ; a minimal upload of 30% of days overall of data would favour retaining this treatment arm in a larger trial
5. To assess the proportion of participants in each intervention arm who complete final evaluation procedures (loss to follow-up rates); a minimum retention of 75% of participants enrolled would favour execution of a larger clinical trial

DESIGN Lawson ACTIVE PATIENT has a 2X2 factorial design. All participants will have access to the information and motivational resource bank, housed on a dedicated study website. Each participant will be randomized (1) to an ePlatform yes/no strategy and (2) to a health coach yes/no strategy. Therefore, some participants will have access to the website only, others to the website & ePlatform, others to the website & coach, and some to the website, ePlatform & coach. By interviewing and surveying participants in each of these groups, the investigators will be able to ascertain if there are components that are redundant or synergistic.

RESOURCE BANK The website sections include (1) 'About' with an overview about GDM, its management, and its complications; (2) 'Perspectives' with video and audio clips and interviews with mothers with a GDM history, physicians, dietitians, and kinesiologists, all describing their experiences living with or managing GDM and highlighting the importance of attending to this condition both during pregnancy and thereafter; (3) 'Nutrition' with descriptions and discussion of impact of eating on glucose control, illustration of the 'healthy plate' concepts, grocery shopping tips, links to healthy recipe banks, a photographic repository of health snack ideas, healthy lunches, and healthy breakfasts; (4) 'Activity' with explanations for pedometer use, step count targets, physical activity targets, step and physical activity monitoring, links to exercise video clips, precautions during pregnancy; and (5) 'Postpartum' which will include future diabetes risk facts relevant to mothers, fathers, and children; diabetes prevention approaches; and planning for future pregnancies.

ePLATFORM WITH SENSORS Participants randomized to the ePlatform strategy (i.e., 50% of participants) will receive a digital scale, physical activity monitor (pedometer), and ePlatform log-in information. They will track daily weights and step counts. They will receive prompts to access educational and motivational tools based on the data that they enter and whether or not they enter data. The investigators will use the ePlatform developed by StepsCount, a Canadian pedometer company with a well-developed ePlatform for pedometer data upload, tracking, and automated messaging. The company is permitting us further customization for study purposes. Participants randomized to the use of an ePlatform in combination with a pedometer and digital scale will have data uploaded onto a secure cloud-based platform controlled by the pedometer and digital scale companies.

HEALTH PROFESSIONAL COACH Participants randomized to the health coach strategy (i.e., 50% of participants) will work by telephone and email with a health coach. The coach will be a health professional hired through the study (dietitian/kinesiologist/nurse). On a weekly basis, She/he will contact the participant to discuss progress and challenges in terms of achieving physical activity goals, rate of GWG, and maintaining health eating patterns. She/he will respond to specific questions on strategies and interplay between health behaviours and parameters such as blood glucose and blood pressure levels. She/he may enquire about any problems associated with higher physical activity levels such as contractions or lower blood sugar levels, and will advise participants accordingly and consult with the treating physician. Participants not randomized to a coaching strategy will be advised to consult with their treating healthcare team directly if they develop symptoms of concern.

Fifty percent of participants will be randomized to a health coach. In turn, half of these participants will also be randomized to the ePlatform with sensors strategy. The health coaching approach will slightly differ between those randomized to the health coach & ePlatform with biosensors strategy vs. those randomized to the health coach without ePlatform strategy.

For those randomized to the health coach & ePlatform with biosensors strategy, the health coach will have access to the data on the ePlatform. This data transfer is termed facilitated relay, the exchange of patient collected health data between patients and providers outside of traditional clinic visits (i.e., electronic and web-based sharing).

Participants randomized to both the ePlatform and the health coach will receive telephone calls from the research assistant/health coach if they are off target despite the platform tools and support. They will be encouraged to consult the resource bank and will brainstorm with the health coach to decide how to achieve their GWG and step count targets.

Participants randomized to the health coach without the ePlatform will receive weekly calls from the health coach, encouraging them to engage in healthy eating practices and aim to achieve the GWG targets recommended by the Institute of Medicine (IOM). They will be encouraged to track their weight gain and physical activity (e.g., walks, gym sessions, classes, activity lists, etc.) and to share this information with the health coach for discussion. However, they will not have access to the study ePlatform and will not be provided with pedometers or digital scales.

At least one coach will be trained for each of the recruitment sites (5). The training will consist of completion of 5 30-minute on-line modules supplemented by teleconferences with our team of experts in health behaviour change (J Fowles, C Shields, C Chan, A-S Brazeau, D Da Costa, K Dasgupta). The on-line training modules for health coaches address motivational communication, key content areas (GDM, health behaviours, stress management), review the bank of resources, discusses the decision trees/algorithms that will create triggers and alerts, and demonstrates navigation of the ePlatform.

SETTING GDM clinics in Montreal (McGill University Health Centre/MUHC with Dr Sara Meltzer, Dr Natasha Garfield, and Dr Rachel Bond; and Centre hospitalier de l'Université de Montréal/CHUM with Dr Ariane Godbout and colleagues), Toronto (Sunnybrook Health Sciences Centre with Dr Illana Halparin, Dr Baiju Shah, and colleagues), Calgary (Rockyview General Hospital with Dr Sonia Butalia and colleagues), Winnipeg (Health Sciences Centre Winnipeg with Dr P Katz and colleagues), and Halifax (Queen Elizabeth II Health Sciences Centre with Dr Tom Ransom and colleagues).

RECRUITMENT GDM clinic staff will invite potentially eligible patients to consider participation. With their permission, contact information will be forwarded to the local ACTIVE PATIENT GDM research assistant. She/he will communicate with the participant to review study procedures and obtain informed consent through an on-line form and telephone conversation. The investigators aim to recruit and enroll at least 5 participants per month per site.

ELIGIBILITY CRITERIA See relevant section

RUN-IN PHASE AND RANDOMIZATION Participants will receive instructions to log onto an electronic platform. This will allow them to view a brief video on GDM-related complications. If the participant logs onto the system within a week of baseline assessment, web-based randomization will be performed. The participant will be encouraged to call or email the research assistant if there is difficulty logging on.

DATA COLLECTION See outcomes for baseline and final data collected

SAMPLE SIZE The investigators will recruit 225 participants across 5 cities, resulting in up to 45 participants per city over 9 months (to allow for 3 month intervention periods) or 5 participants per city per month. The present study is not designed to assess for between-arm differences in GWG or LGA status of the offspring. The intent is to gather experience with logistical procedures, participant perspectives, and estimates of indicators of feasibility.

INCENTIVES On three occasions (completion of the questionnaire at the beginning of the study, completion of the questionnaire and interview before delivery, and completion of the questionnaire and interview 12 weeks after delivery), participants will receive a $20 gift card.

ELIGIBILITY:
Inclusion Criteria:

* Followed by a ACTIVE patient GDM collaborating doctor
* Currently diagnosed with gestational diabetes
* At 20 to <32 weeks during pregnancy
* Conversant in either English or French
* Have frequent access to a Smartphone (iPhone iOS 10.0 or Android version 5.0 or higher) with WIFI capabilities

Exclusion Criteria:

* History or diagnosis of diabetes type 1 or 2
* Currently pregnant with more than one child
* Planning to give birth at a place other than the hospital
* Smokers
* Conditions that are absolute contraindications for exercise during pregnancy (Restrictive lung disease, ruptured membranes, pre-eclampsia, pregnancy-induced hypertension, Premature labour during current pregnancy, persistent bleeding, incomplete cervix, placenta previa, Hemodynamically significant heart disease)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is looking at the effects of interventions on pregnant women with gestational diabetes
Enrollment: 227 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Recruitment | 1 year
  Proportion of candidates with GDM who accept to participate in the study

SECONDARY OUTCOMES:
Use of resource bank | 12 weeks
  Log-ins per participant
Perceived utility of resource bank | 12 weeks
  Post intervention interview. a) What did the participant like about the website resources? b) What did the participant not like about the website? c) Prompts- Did the participant have difficulty logging on? Did the participant have difficulty navigating the site? Did the participant understand the information provided? Did the resource help to motivate the participant?
Step count data | 12 weeks
  Percent of days step count data uploaded in ePlatform arm
Digital weight data | 12 weeks
  Percent of days weight data uploaded in ePlatform arm
Perceived utility of step count monitoring with ePlatform support | 12 weeks
  Post intervention interview. a) Did the participant find it useful to track her step counts? What was useful about it? b) Did the participant find it burdensome to track her step counts? What was burdensome about it? e) Was it easy or was it difficult to use the ePlatform to upload data and review steps and weights? f) Did the participant like the messages from the ePlatform or were they an annoyance? g) Did the participant have any difficulties using a pedometer?
Perceived utility of weight monitoring with ePlatform support | 12 weeks
  Postintervention interview. c) Did the participant find it useful to track her weight? Why? d) Did the participant find it burdensome to track her weight? Why? e) Was it easy or was it difficult to use the ePlatform to upload data and review steps and weights? h) Did the participant have any difficulties using the digital scale?
Number of planned weekly conversations completed with health coach | 12 weeks
  Percent of weeks with health coach contact
Perceived utility of health coaching conversations | 12 weeks
  Postintervention interview. a) Did the participant find it useful to have a health coach? What was useful about it? b) Was it burdensome to have a health coach? What was burdensome? c) Prompts- Was it easy to find a time to speak with the coach? Were the conversations long enough? Were the conversations too long? What did the participant talk about? Was the information useful? Did the participant feel more motivated by having these conversations?
Completion of evaluation procedures | 12 weeks
  Evaluation metrics will be obtained through in-clinic assessments, on-line questionnaires, chart review, and telephone/Skype-based interviews.

OTHER OUTCOMES:
Change in physical activity | 12 weeks
  Objective physical activity assessment. At baseline, all participants will be asked to wear a pedometer Piezo Rx(D) with concealed window for a 1-week period.The pedometer will be mailed to the site research assistant in the mailed and stamped envelope provided with an unused pedometer to correct for steps registered during mailing. At two to three weeks before the expected date of delivery or planned date of C-section or 36 weeks' gestation (whichever is first), the 1-week measurement procedure will be repeated. If the participant was in a group that was asked to use a pedometer during the study, she will not need to wear the pedometer with a tamper-proof seal. The participant will continue to use their usual pedometer.
Gestational weight gain (GWG) | 12 weeks
  All prenatal visit weights will be recorded from the medical paper or electronic chart or entered directly onto our data collection forms by the research assistant or collaborating physician. Participants will be weighed at all clinic visits by the research assistant or collaborating physician. GWG per week will be calculated.
Blood pressure | 12 weeks
  Blood pressure will be assessed at clinic visits by the research assistant or collaborating physician. From 6 automated measurements, the latter 5 systolic and diastolic measures will be separately averaged
Glucose levels | 12 weeks
  Mean glucose levels (before and after meals, at bedtime) will be abstracted at each clinic visit based on participant records
Content of conversations with health coach | 12 weeks
  Health coaches will maintain a log of communications with study participants to allow us to ascertain the frequency and nature of communications as well as the overall time required.
Offspring birthweight percentile | at birth
  Chart review. Offspring birthweight, length, sex. Will be used to classify as large, small, or appropriate for gestational age
Gestational age at birth | at birth
  Chart review
Delivery method | at birth
  Chart review.
Apgar score | at birth
  Chart review
Completion of postpartum screen for diabetes | 12 weeks' postpartum
  Completion of oral glucose tolerance testing. Ascertained by phone interview at 12 weeks' postpartum
Breastfeeding | 12 weeks' postpartum
  Ascertained by phone interview. Between the birth of the participant's baby and now, how have has the participant been feeding her baby?
  * Breastfeeding alone: Specify number of weeks or days
  * Formula feeding alone: Specify number of weeks or days
  * Mix of the two: Specify number of weeks or days

CONTACTS AND LOCATIONS:
Overall Officials: Kaberi Dasgupta, MD, MSC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (6):
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - IWK Helath Centre, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Background] Dasgupta K, Chan D, Bond R, Wang SJ, Garfield N, Coolen J, Halperin IJ, Peters TM, Shen GX, Yamamoto J, Butalia S, Dowling J, Rendon L, Haichin K, Sharafi M, Shields C, Godbout A, Costa DD, Kaouache M, Shah BR, Rahme E, Brazeau AS, Meltzer S; ACTIVE PATIENT GDM team. Step and weight tracking with targets and coaching interventions in gestational diabetes: A randomized factorial feasibility trial. Diabetes Res Clin Pract. 2025 Jun;224:112241. doi: 10.1016/j.diabres.2025.112241. Epub 2025 May 9. PMID 40349846